CLINICAL TRIAL: NCT00192972
Title: A Randomized Trial of the Ostial Versus the Extra-Ostial Ablation Strategy for Atrial Fibrillation (LASso Vs CARto)
Brief Title: A Randomized Trial of the Ostial Versus the Extra-Ostial Ablation Strategy for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Medtronic (Industry); Biosense Webster, Inc. (Industry); Abbott Medical Devices (Industry); Guidant Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: LASCAR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-12-22 (Estimated); Status verified 2003-11

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Catheter ablation; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

INTERVENTIONS:
Procedure: Catheter ablation (pulmonary vein isolation)

SUMMARY:
Both segmental, ostial and circumferential, extra-ostial pulmonary vein (PV) isolation have been proven effective in the treatment of atrial fibrillation.

In this study patients with symptomatic paroxystic or persistent AF were randomised to one of the above mentioned ablation methods. The primary endpoints were recurrent AF and recurrence of left atrium-PV conduction.

DETAILED DESCRIPTION:
Both segmental, ostial and circumferential, extra-ostial pulmonary vein (PV) isolation have been proven effective in the treatment of atrial fibrillation.

In this study with symptomativ paroxystic or persistent AF were randomised to one of the above mentioned ablation methods. Each patient was allowed a maximum of two ablation procedures. Holter monitoring for 14-days periods will be performed at 3 months after ablation. The patiens are seen at out-patient visits at 1, 3, 6, 9, and 12 months after the ablation procedure.

Primary endpoints were recurrent AF and recurrence of left atrium-PV conduction.

Secondary endpoints were:

* safety
* resumption of LA-PV conduction
* alterations in neurohormones
* socio-economics aspects(cost effectiveness)
* changes in inflammatory markers
* quality of life
* alterations in signal averaged P wawe signals
* evaluation of the predictive value of these variables to predict recurrence of AF

ELIGIBILITY:
Inclusion Criteria:

* symptomatic paroxysmal or persistent AF for more than 6 months, with at least 3 episodes in 3 months and with insufficient effect of at least 2 pharmacological regimens

Exclusion Criteria:

* congenital heart disease
* age under 18 years
* significant valve disease
* left atrial size > 55 mm
* prior ablation for AF
* Severe heart failure (LVEF < 20 % and/or NYHA class IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-11; Study Completion 2005-06

PRIMARY OUTCOMES:
overall efficacy (= freedom from symptomatic, ECG documented AF or organized LA tachycardia (with a duration of > 10 min) without receiving antiarrhythmic medication)

SECONDARY OUTCOMES:
- safety
- resumption of LA-PV conduction
- neurohormones
- socio-economics (cost effectiveness)
- inflammatory markers
- quality of life
- signal averaged P wave signals-

CONTACTS AND LOCATIONS:
Overall Officials: Brian Nilsson, MD, Principal Investigator — Rigshospitalet, Denmark; Xu Chen, MD, Principal Investigator — Righospitalet, Copenhagen, Denmark; Steen M Pehrson, MD, Principal Investigator — Righospitalet, Copenhagen, Denmark; Lars Køber, MD, Principal Investigator — Righospitalet, Copenhagen, Denmark; Jørgen Hilden, MD, Principal Investigator — Department of biostatistics, University of Copenhagen; Jesper H Svendsen, MD, Principal Investigator — Righospitalet, Copenhagen, Denmark
Locations (1):
- Righospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Oral H, Chugh A, Lemola K, Cheung P, Hall B, Good E, Han J, Tamirisa K, Bogun F, Pelosi F Jr, Morady F. Noninducibility of atrial fibrillation as an end point of left atrial circumferential ablation for paroxysmal atrial fibrillation: a randomized study. Circulation. 2004 Nov 2;110(18):2797-801. doi: 10.1161/01.CIR.0000146786.87037.26. Epub 2004 Oct 25. PMID 15505091